CLINICAL TRIAL: NCT07239765
Title: An Open-label Study to Evaluate the Safety, Efficacy, and Population Pharmacokinetic Characteristics of Amphotericin B Cholesteryl Sulfate Complex Injection in Patients With Invasive Mold Disease
Brief Title: A Study to Evaluate the Safety, Efficacy, and PPK of ABCD in Patients With IMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LXMSB201902/PRO-III
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Invasive Mold Disease

STUDY DESIGN:
Intervention Model Description: Multicenter, Open-label, Single-arm Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABCD (Experimental): Patients received ABCD at a dose of 3-4 mg/kg for 2-12weeks
  Interventions: Drug: ABCD

INTERVENTIONS:
Drug: ABCD — intravenous infusion

SUMMARY:
Amphotericin B Cholesteryl Sulfate Complex (ABCD) is a generic drug of amphotericin B colloidal dispersion. This study aimed to explore the safety and efficacy of ABCD in patients with invasive mold disease.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age;
* Participant had a diagnosis of proven/probable invasive mold disease (IMD) as determined according to European Organization for Research and Treatment of Cancer/Mycoses Study Group (EORTC-MSG) criteria (2019 version) or proven/probable talaromycosis as determined according to diagnostic criteria for endemic mycosis.

Exclusion Criteria:

* Allergy to amphotericin B or cholesteryl sulfate complex;
* Mycoses only involved skin above fascia;
* Expected survival less than 2 months;
* Pregnant or breast-feeding;
* Non-negative result on HIV antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Up to 14 weeks

SECONDARY OUTCOMES:
The percentages of the patients who completed the 2 week ABCD therapeutic regimen | Up to 12 weeks
The percentages of the patients who completed the 4 week ABCD therapeutic regimen | Up to 12 weeks
The percentages of the patients who completed the 6 week ABCD therapeutic regimen | Up to 12 weeks
The proportion of patients achieving the clinical response of complete remission (CR), partial remission (PR) or stable disease (SD) | Up to 12 weeks
The proportion of patients achieving the clinical response of CR or PR | Up to 12 weeks
The proportion of patients with a microbiological response of eradication or presumed eradication | Up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital Of Guangzhou Medical University, Guangzhou, China